CLINICAL TRIAL: NCT04631510
Title: A Pilot Study of Gabapentin for Sleep in Critically Ill Patients
Brief Title: Gabapentin for Sleep in Critically Ill Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13560
Record Dates: First submitted 2019-12-03; First posted 2020-11-17 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Intensive Care Unit Sleep Disruption
Keywords: Sleep disruption; intensive care unit; gabapentin
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Critically ill patients (Experimental): Administer gabapentin 300 mg PO at 8 PM for sleep
  Interventions: Drug: Gabapentin 300 mg PO at 8 PM

INTERVENTIONS:
Drug: Gabapentin 300 mg PO at 8 PM — Administer gabapentin 300 mg PO at 8 PM for sleep

SUMMARY:
Sleep disruption in the intensive care unit (ICU) is a common comorbidity associated with patient morbidity and distress. There are no recommended pharmacologic interventions for sleep promotion, and many pharmacologic solutions may actually increase the risk of adverse outcomes rather than impart benefits. Gabapentin, an anticonvulsant with applications in neuropathic pain, has been investigated for sleep promotion in various populations of outpatients. Here investigators propose a pilot study of gabapentin as a therapy for sleep disruption in the ICU. Outcomes measured will be sleep quality as measured by RCSQ (Richards-Campbell Sleep Questionnaire), wrist actigraphy, EEG, and BIS monitoring. The goal is to enroll 80 critically ill patients, 40 intubated and 40 non-intubated patients. The study will take place over 2 nights, with baseline sleep measurements occurring on the first night and gabapentin administration with repeat sleep measurements on the second night.

DETAILED DESCRIPTION:
Sleep disruption in the intensive care unit (ICU) is a common comorbidity. In addition to being a source of emotional distress for many patients, sleep disturbance may be associated with ICU delirium, prolonged need for respiratory support, and immune and neurocognitive dysfunction. Since sleep is a potentially modifiable risk factor for ICU outcomes, there has been increased interest in sleep study and promotion in critically ill patients, as evidenced by the inclusion of sleep disruption in the 2018 Society of Critical Care Medicine Clinical Practice Guidelines. Although these Guidelines make soft recommendations for non-pharmacologic strategies to improve sleep in this patient population, these strategies are often lacking in efficacy and/or evidence. There are no recommended pharmacologic interventions for sleep promotion, and many pharmacologic solutions may actually increase the risk of adverse outcomes rather than impart benefits.

Gabapentin, an anticonvulsant with applications in neuropathic pain, has been investigated for sleep promotion in various populations of outpatients. In non-ICU patients, gabapentin is an effective therapy for insomnia in patients with restless leg syndrome or chronic neuropathy. Even in patients without these comorbidities, gabapentin has shown efficacy compared with placebo in improving sleep duration and depth. Gabapentin has several advantages compared to common sedatives used in the ICU, including no increased day drowsiness, no QTc prolongation, and some studies suggesting no association with delirium, particularly when used in a daily dose < 600 mg. Although caution must be used in dosing this drug in patients with renal dysfunction, a dose of up to 300 mg daily may be used if CrCl < 15 ml/m, and doses of up to 300 mg after hemodialysis (HD) have been used safely in patients with end stage renal disease (ESRD). Additionally, its generic status and broad therapeutic index make it a cost-effective and attractive agent for further study and use.

Here investigators propose a pilot study of gabapentin as a therapy for sleep disruption in the ICU. To date, there have been no studies of gabapentin use for sleep in the ICU; this study would represent the first of its kind. Given the magnitude of the problem represented by sleep disruption in the ICU, the ability of gabapentin to mitigate insomnia in outpatients, and the low side effect profile and wide therapeutic window of gabapentin, studying the effects of gabapentin on sleep disruption in the ICU is a logical and potentially practice changing step.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the ICU or step-down unit (neurologic intermediate care center or Pratt 8) for ≥ 24 hours
2. ≥ 1 risk factor for delirium: benzodiazepine use, blood transfusions, age >60 years, dementia, prior coma, pre-ICU emergency surgery or trauma, American Society of Anesthesia (ASA) score > 3, Acute Physiology and Chronic Health Evaluation II (APACHE II) >12, admission because of a neurologic disease, trauma, and the use of psychoactive medication (e.g., antipsychotics, anticonvulsants)
3. Age ≥ 18 years old
4. Anticipated ICU or step-down unit length of stay ≥ 48 hours past time of enrollment
5. Riker score goal of 3 or 4

Exclusion Criteria:

1. Pregnant women
2. Age < 18 years old
3. Wards of the state or prisoners
4. Patients who were considered by their primary physician to be too unstable to undergo this investigation
5. Comatose patients or patients with severe debilitating neurologic disease such as cerebrovascular accidents, intracranial hemorrhage, subdural hematoma, intracranial primary or secondary cancers, or anoxic-hypoxic encephalopathy
6. Moribund patient expected to die within 24 hours
7. Expected change in intubation status within 24 hours of enrollment
8. Gabapentin or pregabalin use in the last 7 days or at baseline
9. Patients with a known sensitivity to gabapentin
10. Currently receiving a non-benzodiazepine hypnotic (i.e. zolpidem, eszopiclone)
11. Need for every hour neurologic checks
12. Creatinine clearance < 15ml/min or need for renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
change in sleep efficiency | for 12 hours after gabapentin administration
  improvement in sleep efficiency index (SEI) over baseline as measured by Richards-Campbell Sleep Questionnaire (RCSQ)

SECONDARY OUTCOMES:
change in sleep quality: total sleep duration/time (TST) | for 12 hours after gabapentin administration
  BIS monitoring for total sleep duration/time (TST)
change in sleep quality: sleep latency | for 12 hours after gabapentin administration
  Sleep efficiency (TST/TRT), sleep latency
change in sleep quality: REM latency | for 12 hours after gabapentin administration
  REM latency
change in sleep quality | for 12 hours after gabapentin administration
  wakefulness after sleep onset (WASO)
sleep quality: number of awakenings/arousals (#arousals/hour) | for 12 hours after gabapentin administration
  number of awakenings/arousals (#arousals/hour)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Tsai, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No